CLINICAL TRIAL: NCT02672371
Title: The Effects of Sensory Training On Pain Modulation, Cognition and Time to Fatigue in Healthy Adults
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was not approved for the IRB; we then had no funds to reapply
Sponsor: Spaulding Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Felipe Fregni, Principal Investigator, Spaulding Rehabilitation Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 2015P002574
Record Dates: First submitted 2015-12-08; First posted 2016-02-03 (Estimated); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Healthy Participants

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active eMNS (Experimental): Subjects with receive active eMNS for 20 minutes.
  Interventions: Device: Active eMNS
- sham eMNS (Sham Comparator): Subjects with receive sham eMNS for 20 minutes.
  Interventions: Device: Sham eMNS

INTERVENTIONS:
Device: Active eMNS — Each session will consist of right eMNS stimulation that will last 20-minutes. The frequency of stimulation will be random assigned using random frequency interval. The electrodes that will be used will be standard transcutaneous electrodes. The electrodes will be placed on the wrist.
  Arms: active eMNS
Device: Sham eMNS — Each session of sham eMNS will be the same as active, except the device will be turned off. Similar parameters will be used (for 20 minutes and same electrode placement), except no stimulation will be delivered.
  Arms: sham eMNS

SUMMARY:
The study is a randomized clinical trial that is assessing the effects of sensory training on pain modulation, cognition, and physical endurance (time to fatigue) in healthy participants

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent to participate in the study
* Able to perform physical activities such as cycling
* 18-40 years old
* BMI<27
* Practice of moderate intensity aerobic physical activity less than 150 minutes per week

Exclusion Criteria:

* Hypertension
* Diabetes
* Cardiovascular disease
* Subjects with pacemakers, and/or implantable cardioverter-defibrillators
* History of asthma with active symptomatology in the past year, pulmonary disease or use of inhalers
* Physical disability, neurological and/or psychological disorder that precludes safe and adequate testing
* Conditions that may impair the ability to feel pain
* Mental impairment with limited ability to cooperate
* Uncorrected medical conditions, such as significant anemia, important electrolyte imbalance, or hyperthyroidism
* Pregnancy or trying to become pregnant in the next 6 months
* History of alcohol or drug abuse within the past 6 months as self-reported
* Epilepsy
* Suffering from severe depression (with a score >30 in the Beck Depression Inventory)
* History of unexplained fainting spells as self-reported
* Head injury resulting in more than a momentary loss of consciousness
* History of neurosurgery as self-reported
* Use of antiepileptic and/or hypnotic medications like carbamazepine, valproate acid, gabapentin, zolpidem, etc.
* Use of medication with potential cardiovascular influence
* Active smoker, or history of smoking in the last 6 months
* Skin lesion or open wounds around or in area of electrode application
* Tattoos in upper limb or along the nerve tract

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2017-06 (Estimated); Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
PPT | Between Visit 2 and 3...where Visit 1 = baseline, Visit 2 = stimulation visit, randomly assigned sham or active (about 2 days from baseline), and Visit 3 = other stimulation visit, sham or active - one not received before (about 1 week from visit 2)
  Pain threshold as measured by Pressure Pain Threshold (PPT) between Visits 2 and 3 (active stimulation and sham, order randomized).
DNIC | Between Visit 2 and 3...where Visit 1 = baseline, Visit 2 = stimulation visit, randomly assigned sham or active (about 2 days from baseline), and Visit 3 = other stimulation visit, sham or active - one not received before (about 1 week from visit 2)
  Pain threshold as measured by Descending Noxious Inhibitory Control (DNIC) between Visits 2 and 3
VAS | Between Visit 2 and 3...where Visit 1 = baseline, Visit 2 = stimulation visit, randomly assigned sham or active (about 2 days from baseline), and Visit 3 = other stimulation visit, sham or active - one not received before (about 1 week from visit 2)
  Pain threshold as measured by Visual Analogue Scale (VAS) between Visits 2 and 3

SECONDARY OUTCOMES:
EEG | Visit 2 and Vist 3...where Visit 1 = baseline, Visit 2 = stimulation visit, sham or active (about 2 days from baseline), and Visit 3 = stimulation visit, sham or active (about 1 week from visit 2)
  Spontaneous oscillatory brain activity as measured by EEG using a wireless Enobio system (Neuroelectrics, Barcelona, Spain).
Attention Task | Visit 2 and 3...where Visit 1 = baseline, Visit 2 = stimulation visit, randomly assigned sham or active (about 2 days from baseline), and Visit 3 = other stimulation visit, sham or active - one not received before (about 1 week from visit 2)
  Cognitive Performance (for attention) as measured by the Attention Network Task
N Back test | Visit 2 and 3...where Visit 1 = baseline, Visit 2 = stimulation visit, randomly assigned sham or active (about 2 days from baseline), and Visit 3 = other stimulation visit, sham or active - one not received before (about 1 week from visit 2)
  Cognitive Performance (for working memory) as measured by the
Time to fatigue | Visit 2 and 3...where Visit 1 = baseline, Visit 2 = stimulation visit, randomly assigned sham or active (about 2 days from baseline), and Visit 3 = other stimulation visit, sham or active - one not received before (about 1 week from visit 2)
  Time to fatigue as measured by total cycling time at 80% of peak power.
Perception of physical exertion | Visit 1, 2, and 3...where Visit 1 = baseline, Visit 2 = stimulation visit, randomly assigned sham or active (about 2 days from baseline), and Visit 3 = other stimulation visit, sham or active - one not received before (about 1 week from visit 2)
  Perception of physical exertion as measured by the 6-20 Borg Scale
Heart rate | Visit 1, 2, and 3...where Visit 1 = baseline, Visit 2 = stimulation visit, randomly assigned sham or active (about 2 days from baseline), and Visit 3 = other stimulation visit, sham or active - one not received before (about 1 week from visit 2)
  Heart rate as measured by a standard electrocardiogram
Respiratory rate | Visit 1, 2, and 3...where Visit 1 = baseline, Visit 2 = stimulation visit, randomly assigned sham or active (about 2 days from baseline), and Visit 3 = other stimulation visit, sham or active - one not received before (about 1 week from visit 2)
  Respiratory rate as measured by a belt transducer

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Fregni, MD, PhD, MPH, Principal Investigator — Spaulding Rehabilitation Hospital
Locations (1):
- Spaulding Rehabilitation Network Research Institute, Charlestown, Massachusetts, United States